CLINICAL TRIAL: NCT06055166
Title: A Prospective, Multi-cohort, Single-center Phase II Clinical Study of Chemoradiotherapy Sequential Fluzoparib in Pan-solid Tumors
Brief Title: A Clinical Study of Chemoradiotherapy Sequential Fluzoparib in Pan-solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ChongqingCancer CZLS2023154-A
Record Dates: First submitted 2023-07-26; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-07

CONDITIONS: PARP Inhibitor for Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — fluzoparib; Capecitabine

STUDY DESIGN:
Intervention Model Description: 4 arms include rectal cancer, non-small cell lung cancer, oesophageal squamous cancer, and cervical cancer, accept sequential fluzoparib after chemoradiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- untreated surgically resectable rectal cancer (Experimental)
  Interventions: Drug: Fluzoparib monotherapy or Fluzoparib with Camrelizumab(Only non-small cell lung cancer arm) ,or Fluzoparib combined with capecitabine (only rectal cancer arm))
- untreated locally advanced unresectable non-small cell lung cancer (Experimental)
  Interventions: Drug: Fluzoparib monotherapy or Fluzoparib with Camrelizumab(Only non-small cell lung cancer arm) ,or Fluzoparib combined with capecitabine (only rectal cancer arm))
- untreated locally advanced unresectable esophageal squamous cell carcinoma (Experimental)
  Interventions: Drug: Fluzoparib monotherapy or Fluzoparib with Camrelizumab(Only non-small cell lung cancer arm) ,or Fluzoparib combined with capecitabine (only rectal cancer arm))
- untreated locally advanced unresectable cervical carcinoma (Experimental)
  Interventions: Drug: Fluzoparib monotherapy or Fluzoparib with Camrelizumab(Only non-small cell lung cancer arm) ,or Fluzoparib combined with capecitabine (only rectal cancer arm))

INTERVENTIONS:
Drug: Fluzoparib monotherapy or Fluzoparib with Camrelizumab(Only non-small cell lung cancer arm) ,or Fluzoparib combined with capecitabine (only rectal cancer arm)) — Arm A: untreated surgically resectable rectal cancer. Patients accept preoperative long-range synchronous chemoradiotherapy → fluzoparib combined with capecitabine (Q3W, 4 treatment cycles) → surgery → observation and follow-up Arm B, C and D: include untreated locally advanced unresectable non-small cell lung cancer, esophageal squamous cell carcinoma and cervical carcinoma. Patients accept radical synchronous chemoradiotherapy following → fluzoparib combined with camrelizumab or fluzoparib monotherapy maintenance treatment for 17 cycles

SUMMARY:
This study is a prospective, multi-cohort, single-centre, phase II clinical trial designed to initially explore the efficacy and safety of sequential fluzoparib with chemoradiotherapy in pan-solid tumours. The study is designed for patients with untreated surgically resectable rectal cancer and untreated locally advanced unresectable non-small cell lung cancer, oesophageal squamous cancer, and cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

-

Subjects must meet all of the following criteria to be enrolled in this study:

1. subjects voluntarily enrolled in this study, signed informed consent, good compliance, and co-operated with follow-up visits;
2. age 18-75 years (calculated on the date of signing the informed consent);
3. histologically or cytologically confirmed solid tumours as follows: Cohort A: patients with resectable locally advanced rectal adenocarcinoma not previously treated for rectal cancer (clinical stage T3-4 or N+ as assessed by MRI, according to AJCC 8th edition staging), with the lower edge of the tumour ≤ 10 cm away from the anal verge, with R0 resection predicted and planned for surgery after neoadjuvant therapy, and with no contraindications to surgery; Cohort B: patients with locally advanced, unresectable NSCLC with histologically or cytologically confirmed diagnosis who have not previously received treatment for lung cancer (IIIA, IIIB, IIIC, according to the International Manual of Thoracic Oncology Lung Cancer Staging Studies 8th edition staging); Cohort C: patients with locally advanced, unresectable or contraindicated for or refusing surgery for squamous oesophageal cancer with histological or cytological confirmation who had not received previous treatment for oesophageal cancer (clinical staging T1b-4bN0M0/T1-4bN+M0, according to AJCC 8th edition staging); Cohort D: Cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix that has not received prior treatment for cervical cancer (excluding surgical pathological staging) and that has been confirmed by pathohistology. Clinical staging or imaging staging or surgical pathological staging of locally advanced cervical cancer (2018 FIGO staging of IB3, Stage IIA2-IVA patients);
4. NSCLC without sensitive EGFR, ALK or ROS1 gene mutations confirmed by histological or cytological specimens;
5. ECOG PS score: 0 to 1;
6. subjects with normal swallowing function;
7. normal major organ function, including:

   a) Routine blood tests (no transfusion of blood or blood products, no correction with G-CSF and other haematopoietic stimulating factors within 14 days prior to the first treatment): i. Neutrophil count ≥ 1.5 × 109/L ii. Platelet count ≥ 100×109/L iii. Haemoglobin ≥ 90 g/L. b) Blood biochemistry: i. Total bilirubin ≤ 1.5×ULN ii. ALT ≤ 2.5×ULN, AST ≤ 2.5×ULN. iii. iii. serum creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min c) Coagulation function: i. International Normalised Ratio (INR) ≤ 1.5 x ULN ii. Activated partial thromboplastin time (APTT) ≤ 1.5 x ULN
8. Female subjects of childbearing potential are required to have a negative serum pregnancy test within 72 hours prior to the first dose and are not breastfeeding and are using effective contraception (e.g., IUD, birth control pills, or condoms) for the duration of the trial, and for 6 months after the last administration of fluzoparib/chemotherapy, or 2 months after the last administration of karelizumab, whichever is longer; for male subjects whose partner is a female of childbearing potential, the results of the serum pregnancy test must be negative and they must be not breastfeeding. male subjects whose partner is a female of childbearing potential should be surgically sterilised or agree to use effective contraception for the duration of the trial and for 6 months after the last administration of fluzoparib/chemotherapy or 2 months after the last administration of carrelizumab, whichever is longer, and sperm donation is not permitted during the study.
9. patients judged by the investigator to be acceptable for the study intervention programme.

Exclusion Criteria:

* Subjects with any of the following traits or conditions will not be allowed to enter this study:

  1. patients with a previous history of perforation, fistula, bleeding or airway stenosis;
  2. a history of allergy or risk of allergy to the study intervention protocol;
  3. subjects may receive other systemic anti-tumour therapy during the study period;
  4. the presence of abnormal gastrointestinal function which, in the judgement of the investigator, may interfere with drug absorption
  5. the presence of uncontrollable pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
  6. subjects with congenital or acquired immune deficiency (e.g., HIV-infected), or active hepatitis (Hepatitis B reference: HBsAg positive, HBV DNA ≥2000 IU/ml; Hepatitis C reference: HCV antibody positive, HCV viral copy number > upper limit of normal);
  7. have clinical symptoms or diseases of the heart that are not well controlled, such as: (1) NYHA class 2 or higher heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant supraventricular or ventricular arrhythmia that requires treatment or intervention (5) those with a QTc > 470 ms;
  8. those with abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds), bleeding tendency or who are receiving thrombolytic or anticoagulant therapy are permitted to receive low-dose low molecular heparin or oral aspirin for prophylactic anticoagulation during the trial;
  9. have had a serious infection (CTCAE > grade 2) within 4 weeks prior to first use of study drug, such as severe pneumonia requiring hospitalisation, bacteraemia, or infectious co-morbidities; except for prophylactic antibiotic use in those who have baseline chest imaging suggestive of active lung inflammation, signs and symptoms of infection within 14 days prior to the first use of study drug, or who require treatment with oral or intravenous antibiotics ;
  10. patients with any active autoimmune disease or a history of autoimmune disease with potential for relapse [including, but not limited to, autoimmune hepatitis, interstitial pneumonitis, uveitis, enterocolitis, pituitary gland inflammation, vasculitis, nephritis, hyperthyroidism, and hypothyroidism (patients who can be controlled by hormone replacement therapy alone may be enrolled)] are not eligible for enrollment into Cohort B; patients with skin diseases that do not require systemic therapy Patients with skin diseases that do not require systemic treatment, such as leukoplakia, psoriasis, alopecia areata, patients with type I diabetes mellitus controlled by insulin therapy or patients with a history of asthma that has completely resolved in childhood and does not require any intervention can be enrolled; patients with asthma requiring bronchodilator intervention cannot be enrolled in Cohort B;
  11. women who are pregnant or breastfeeding;
  12. the presence of other factors that, in the judgement of the investigator, could lead to forced termination of the study midway, such as the presence of other serious illnesses (including psychiatric illnesses) that require comorbid treatment, alcoholism, drug abuse, family or social factors that may affect the safety of or compliance with the subject;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
pCR | within 14 working days after operation
  Pathological Complete Response
PFS rate | from initially chemoradiotherapy follow up 12 months
  12-month Progression-Free Survival Rate

SECONDARY OUTCOMES:
MPR | within 14 working days after operation
  Main Pathological Remission
R0 resection rate | within 14 working days after operation
  R0 resection rate
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-Free-Survival
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Overall Survival
ORR | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Objective Response Rate
AEs | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  adverse events

IPD SHARING:
Plan to Share IPD: No